CLINICAL TRIAL: NCT07068412
Title: Impact of 3D-Printed Anatomical Models on Patient Understanding, Anxiety, Patient-Doctor Relationship, and Overall Satisfaction During the Informed Consent Process in Orthognathic Surgery: A Randomized Clinical Trial
Brief Title: Impact of 3D-Printed Anatomical Model on Patient Understanding in Orthognathic Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Razan Baabdullah, Assistant professor of oral and maxillofacial surgery Affiliation: King Abdulaziz University, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 139-11-24
Record Dates: First submitted 2025-06-20; First posted 2025-07-16 (Actual); Last update posted 2025-07-16 (Actual); Status verified 2025-07

CONDITIONS: Skeletal Deformities; Orthognathic Surgical Procedures; Anxiety; Patient Education
Keywords: Skeletal deformities; Skeletal class II; Skeletal class III; Orthognathic surgery; Patient understanding; Patients' satisfaction; Patient-doctor relationship; Anxiety level; anatomical models; 3D printed models; Patient education
MeSH Terms: conditions — Anxiety Disorders | interventions — Orthognathic Surgery

STUDY DESIGN:
Intervention Model Description: This single-blinded randomized controlled trial conducted at King Abdulaziz Dental Hospital to evaluate the impact of three dimensional (3D)-printed anatomical models on patient understanding, anxiety, satisfaction, and communication during the informed consent process for orthognathic surgery. Sixty adult patients scheduled for double- or triple-jaw surgery will be randomly assigned to either a control group (two dimensional (2D) imaging and verbal explanation) or an intervention group (2D imaging plus 3D-printed models). Models were created from CBCT scans using 3D Slicer software and printed with Formlabs resin printers. All consultations are standardized and delivered by calibrated surgeons. Validated Arabic questionnaires will be used to assess outcomes.
Who Masked: Outcomes Assessor
Masking Description: Single
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 2D Surgical Simulation (Active Comparator): This group received an orthognathic surgery consultation incorporating two-dimensional images generated from virtual surgical planning. These images illustrated the patient's current skeletal deformity and the anticipated surgical movements, providing a visual aid to enhance understanding and facilitate informed decision-making.
  Interventions: Combination Product: 2D Visual Representations of Skeletal Movements in Orthognathic Surgery
- 3D Surgical Simulation (Experimental): This group received an orthognathic surgery consultation using 3D-printed anatomical models. The models, representing skeletal Class II and Class III deformities, were customized and modified to simulate osteotomies. During the consultation, these models are used to demonstrate the planned surgical movements, providing patients with a tangible, visual understanding of their condition and the proposed treatment.
  Interventions: Combination Product: 3D-printed Orthognathic Surgical Simulation

INTERVENTIONS:
Combination Product: 3D-printed Orthognathic Surgical Simulation — Two standardized 3D-printed anatomical models were created-one representing skeletal Class II and the other skeletal Class III. Simulated osteotomies, including Le Fort I and Bilateral Sagittal Split Osteotomies, were performed on the models to demonstrate surgical movements. These models are used to help patients visualize the procedures planned for their specific cases.
  Other Names: 3d-printed anatomical models
  Arms: 3D Surgical Simulation
Combination Product: 2D Visual Representations of Skeletal Movements in Orthognathic Surgery — Two-dimensional images generated from virtual surgical planning-one depicting a Class II skeletal deformity and the other a Class III malocclusion-are used to illustrate the patient's condition and demonstrate the anticipated surgical movements.
  Arms: 2D Surgical Simulation

SUMMARY:
The goal of this clinical trial is to learn whether using three dimensional (3D)-printed anatomical models improves the informed consent process for participants undergoing orthognathic surgery. The trial also explores how these models affect participants understanding, anxiety, satisfaction, and communication with the surgeon.

The main questions it aims to answer are:

* Do 3D-printed anatomical models improve participants understanding of their jaw condition and the surgical procedure?
* Do they reduce participants anxiety before surgery?
* Do they enhance overall participants satisfaction and the physician-patient relationship?

Researchers compares participants who received standard two dimensional (2D) imaging and verbal explanations with those who received the same information plus 3D-printed jaw models.

Participants:

* Scheduled for double- or triple-jaw orthognathic surgery
* Randomly assigned to receive either traditional 2D education or the 3D-printed model intervention
* Complete a validated questionnaires assessing understanding, anxiety, satisfaction, and doctor-patient communication

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (aged 18 and above)
* Scheduled for orthognathic surgery (specifically double-jaw or triple-jaw procedures)

Exclusion Criteria:

* Pediatric patients (under 18 years old)
* Patients undergoing re-do/revision surgery
* Patients with psychiatric disorders
* Patients receiving only orthodontic treatment
* Patients undergoing single-jaw surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-08-30 (Estimated)

PRIMARY OUTCOMES:
Patient understanding | Baseline
  Patient comprehension scores of their jaw condition, planned surgical procedures (Le Fort I, bilateral sagittal split osteotomy, and genioplasty), potential complications, expected outcomes, and the overall consent process, measured by a structured questionnaire at the time of consent.

SECONDARY OUTCOMES:
Anxiety level | Baseline
  Patient anxiety levels related to orthognathic surgery, as measured by the validated Arabic version of the State-Trait Anxiety Inventory (STAI), a 20-item self-administered questionnaire.
Patient-doctor relationship | Baseline
  Scores for quality of communication and trust between patient and surgeon, as measured by the Arabic version of the Patient-Doctor Relationship Questionnaire (PDRQ-9).
Patient Satisfaction | Baseline
  Patient satisfaction scores regarding the consultation and informed consent process, as measured by the validated Arabic version of the Patient Satisfaction Questionnaire (PSQ-18).

CONTACTS AND LOCATIONS:
Overall Officials: Razan M Baabdullah, BDS,MS,FRCDC, Principal Investigator — King Abdulaziz University, Faculty of Dentistry, Department of Oral and Maxillofacial Surgery
Locations (2):
- Saudi Arabia (2):
  - Razan Baabdullah, Jeddah, Mecca Region
  - King Abdulaziz University Dental Hospital, Jeddah

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2025-06-01): https://cdn.clinicaltrials.gov/large-docs/12/NCT07068412/Prot_SAP_000.pdf